CLINICAL TRIAL: NCT06986980
Title: Intestinal Microsporidiosis in French Heart Transplant Recipients
Brief Title: Intestinal Microsporidiosis in French Heart Transplant Recipients (CARMIC)
Acronym: CARMIC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2025 NOURRISSON GARROUSTE
Record Dates: First submitted 2025-04-17; First posted 2025-05-23 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-04

CONDITIONS: Microsporidiosis Intestinal; Heart Transplant Infection
Keywords: microsporidiosis; Enterocytozoon bieneusi; Encephalitozoon intestinalis; Encephalitozoon hellem; solid organ transplant; heart transplant
MeSH Terms: conditions — Microsporidiosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators propose to carry out a national retrospective study to collect epidemiological, biological, clinical and therapeutic data on microsporidiosis among heart transplant patients.

DETAILED DESCRIPTION:
Microsporidia constitute a large family of intracellular eukaryotes infecting a wide range of hosts, ranging from insects to mammals and birds. Within this group, some species are responsible for intestinal syndromes manifested by abundant watery diarrhea, which can be particularly severe in immunocompromised individuals. In the 1980s, HIV-positive patients at the AIDS stage represented the primary population at risk. Nowadays, the most frequently affected patients among immunocompromised individuals are solid organ transplant recipients, for whom the management of this infection can be challenging. A neglected pathology until a few years ago, epidemiological data describing intestinal microsporidiosis in solid organ transplant recipients are scarce. The invesigators previously published the first data in kidney and liver transplant recipients. Here the investigators propose to carry out a national retrospective study to collect epidemiological, biological, clinical and therapeutic data on heart transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* heart transplant patients diagnosed with intestinal microsporidiosis
* diagnosis made before December 31, 2024 in France (metropolitan France and overseas territories)

Exclusion Criteria:

-patient opposition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Heart transplant patients with microsporidiosis
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Demographic data: age | 1 year
  expressed in years old
Demographic data: sex | 1 year
  choice between: male/female
Time between transplant and microsporidiosis | 1 year
  expressed in days, or years if >365 days
At diagnosis: number of days since the onset of symptoms | 1 year
  expressed in number of days
Weight loss at diagnosis | 1 year
  expressed in kilogram or in percent (compared to usual weight of the patient)
Dosage of immunosuppressants at diagnosis | 1 year
Time to stool negativation | 1 year
  expressed in number of days between onset of treatment and first negative PCR during follow-up
Creatinine level in blood at Day 0 (diagnosis) and Month 3 | 3 months
  expressed in µM
Numeration of cells in blood: platelets, lymphocytes, neutrophils at Day 0 (diagnosis) and Month 3 | 3 months
  expressed in Giga per litre
Gammaglobulins in blood at diagnosis | 1 year
  expressed in gram per litre

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Gabriel Montpied, Clermont-Ferrand, France